CLINICAL TRIAL: NCT00704665
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Recombinant Human Relaxin in the Treatment of Systemic Sclerosis With Diffuse Scleroderma
Brief Title: Recombinant Human Relaxin in the Treatment of Diffuse Scleroderma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: University of California, Los Angeles (Other); Boston University (Other); University of Chicago (Other); UConn Health (Other); Johns Hopkins University (Other); University of Pittsburgh (Other); Medical University of South Carolina (Other); Stanford University (Other); Georgetown University (Other); University of California, San Diego (Other); Wayne State University (Other); University of Colorado, Denver (Other); Medical College of Wisconsin (Other)
Responsible Party: James R. Seibold, UMDNJ
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2773
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2008-06-25 (Estimated); Status verified 2008-06

CONDITIONS: Systemic Sclerosis
Keywords: Diffuse Scleroderma; Skin score
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Relaxin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Relaxin
- A (Experimental): 10ug/kg/day or 25/ug/kg/day
  Interventions: Drug: Relaxin

INTERVENTIONS:
Drug: Relaxin — 10 ug/kg/day or 25 ug/kg/day
  Arms: A
Drug: Relaxin — Placebo
  Arms: 2

SUMMARY:
Relaxin is a naturally occurring protein prduced by the ovary or placenta in pregnancy. It has ani-fibrotic properties. Previous studies have shown that relaxin is safe at concentrations upto 60 times higher than achieved in pregnancy. Study is designed to see if skin improvement and improvement in functional ability can be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 70 years of age with diffuse SSc
* Disease duration 5 years since the onset of the first non-Raynaud sign or symptom
* A baseline modified Rodnan skin score (MRSS) of 20 or greater, or at least 16 if truncal involvement was present.
* Recombinant human relaxin (10 or 25 ug/kg/day), or placebo was administered for 24 weeks as a continuous subcutaneous infusion and there was a follow-up safety visit at week 28.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 1998-12; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
MRSS | baseline, weeks 4,12, and 24

SECONDARY OUTCOMES:
HAQ-DI | baseline, weeks 4, 12, and 24